CLINICAL TRIAL: NCT07010978
Title: R34 Study 2 - Pilot RCT Testing the Effectiveness of RCCs
Brief Title: Towards Testing the Effectiveness of Recovery Community Centers (RCCs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Bettina B. Hoeppner, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P001189; 1R34DA057604-01 (NIH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; moud; medications for opioid use disorder; recovery; recovery community centers
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: remote, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Community Center (RCC) Linkage (Experimental): These participants will be assigned to visit their local recovery community center at least twice, on two different days, within the first month of the study and to report on their RCC visits.
  Interventions: Behavioral: Recovery Community Center Participation
- Enhanced Treatment as Usual (ETAU) (Active Comparator): These participants will be asked to complete any recovery activity of their choosing at least twice, on two different days, within the first month of the study and to report on their chosen recovery activities.
  Interventions: Behavioral: Enhance Treatment as Usual

INTERVENTIONS:
Behavioral: Recovery Community Center Participation — Recovery community centers are brick and mortar buildings that house recovery-oriented organizations, located in the heart of their communities. They act as recovery hubs, offering a variety of recovery support services in house as well as connecting participants to resources in their area. They are peer-led organizations that are open to anyone in early or long-term recovery from substance use and that recognize that there are multiple pathways to recovery. Study participants will be provided with information about their local RCC (including a video link, contact information, a monthly calendar of events, a list of services and activities offered by the RCC, transportation options, etc.) and will be asked to visit the RCC on two different occasions within one month of enrollment.
  Arms: Recovery Community Center (RCC) Linkage
Behavioral: Enhance Treatment as Usual — In this study, the enhanced treatment as usual intervention will encompass providing participants with information about diverse recovery activities (e.g., mutual help group meetings, exercise, job search, recovery coach meetings, etc.) and then to assign participants to complete a recovery activity of their choosing one two different days within one month after enrollment. Participants can do the same activity twice, or different activities on each of the two days assigned.
  Arms: Enhanced Treatment as Usual (ETAU)

SUMMARY:
The goal of this pilot randomized clinical trial is to prepare for a larger randomized clinical trial (RCT) and collect some early data to learn if the intervention can help people who use medications for opioid use disorder (MOUD). The main questions it aims to answer are:

1. Is it feasible to recruit and randomize people to both treatment groups?
2. Does linking people to recovery community centers lead to better recovery outcomes?

Researchers will compare linking people to recovery community centers (RCC) to enhanced treatment as usual to see if recovery outcomes are different.

In one group, participants will learn about their local RCC and will be asked to visit their local RCC on at least two days and write about their experiences. In the other group, participants will learn about different recovery activities, pick any two, and do the activities of their choice on at least two days. They will also be asked to write about their experiences.

People in both groups will answer online survey questions about their recovery outcomes and well-being in five surveys over one year.

DETAILED DESCRIPTION:
The goal of this study is to prepare for a large-scale RCT. The current study is a pilot randomized clinical trial (RCT) comparing RCC linkage vs. enhanced treatment as usual (ETAU). Persons engaged in MOUD clinical care (n=128) at MOUD-providing clinics near RCCs serving Black communities will be recruited nationwide. The aims of this study are:

Aim 1: Determine the number of study participants enrolled per month. This information will be used for planning a subsequent R01, in line with the goals of the R34 mechanism used to fund this study.

Aim 2: Determine the feasibility of the chosen randomization procedures and groups in terms of (a) study enrollment, (b) completion of recovery activity assignments, and (c) completion of follow-up assessments.

Exploratory Aim 3: Estimate the size of treatment group differences on recovery outcomes over time, including on (a) the Substance Use Recovery Evaluator (SURE); (b) the Brief Measure of Recovery (BMR-4; derived from the Substance Abuse and Mental Health Services Administration's (SAMHSA) definition of recovery); (c) Experience Of Support (derived from SAMHSA goals of peer recovery support services); (d) Brief Assessment of Recovery Capital (BARC-10); and (e) self-report of participation in recovery support services.

Of note, this is a community-engaged research project, involving three community partners (i.e., the Detroit Recovery Project (DRP), Northern Ohio Recovery Association (NORA), and Let's Talk Safety (PILLARS)).

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Uses MOUD (at enrollment; participants may stop using MOUD subsequently) to treat OUD
* Receives MOUD from a clinic/pharmacy located within 15 miles of an RCC vetted by our study team, which serves a Black community (i.e., defined as being located in a ZIP code where ≥27% of the residents are Black, as per US Census)
* Is willing and able to engage in study procedures (i.e., online surveys, timeline follow back interview)
* Is willing to be randomized

Exclusion Criteria:

- Has visited a vetted RCC during the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline
  The recruitment rate will be estimated from the number of study participants enrolled per month; this information will be used for planning a subsequent R01, in line with the goals of the R34 mechanism used to fund this study. The recruitment rate will be reported as mean with standard deviation (based on monthly observations) and will be reported descriptively.

SECONDARY OUTCOMES:
Study Withdrawals | 1 month
  Study withdrawals (i.e., participant-initiated withdrawals from the study after they learn about their randomized treatment assignment) will be reported as the number and percent of participants withdrawing.
Completion of Recovery Activities | 1 month
  To assess the completion rate of assigned recovery activities, we will ask participants to report whether they completed (=1) or did not complete (=0) each of the two recovery activities they will schedule with study staff after enrollment. Completion rates will be presented as the number and percent of participants completing the first or second recovery activity, respectively.
Completion of Follow-up Surveys | Baseline, 1, 3, 6, and 12 month
  To assess completion of study assessments, we will check whether participants completed (including partial completions) (=1) or did not complete (=0) follow-up surveys at each assessment time point. Completion rates will be reported as the number and percent of participants completing them.
Completion of Timeline Follow-Back (TLFB) Interviews | Baseline, 1, 3, 6, and 12 months
  As part of assessing completion of study assessments, we will assess whether study participants completed the Timeline Follow-Back (TLFB) interview (=1) or not (=0) at each assessment time point. In the TLFB interviews, we will ask participants to go back through the last 30 days and report on specific recovery or substance use behaviors. For recovery supports, we will ask participants to tell us on which days they used medications for opioid use disorder or visited their local recovery community center. For substance use, we will ask participants about any non-prescribed opioid use, such as heroin or fentanyl, prescription opioids use without having a prescription for them, and any alcohol use. Completion of TLFB interviews will be reported as number and percent of participants completing them at each assessment point.

OTHER OUTCOMES:
The Substance Use Recovery Evaluator (SURE) | Baseline, 1, 3, 6, and 12 months
  The Substance Use Recovery Evaluator (SURE) is a 21-item self-report measure assessing recovery from drug and alcohol dependence. The 21 items ask about five dimensions relevant to recovery, assessed over the previous week: substance use and coping (6 items), self-care (5 items), relationships (4 items), material resources (3 items), and outlook on life (3 items). Each item is unique and non-redundant with other items on the scale. Questions 1-3 are rated on scale from 1 = "Never" to 5 = "Everyday" and questions 4-21 on a scale of 5 = "All the time" to 1 = "None of the time." Total scores can range from 21 to 63, with higher scores indicating better recovery outcomes.
Brief Measure of Recovery (based on SAMHSA's definition of recovery) | Baseline, 1, 3, 6, and 12 months
  This 4-item self-report measure is derived directly from SAMHSA's (Substance Abuse and Mental Health Administration, 2012) working definition of recovery. The items are (1) "I have relationships and social networks that provide support, friendship, love, and hope"; (2) "I have a stable and safe place to live"; (3) "I have the independence, income and resources to participate in society"; and (4) "I have meaningful daily activities, such as a job, school, volunteerism, family care-taking, or creative endeavors." Each item is rated on a 3-point scale (0=no, not at all, 1=yes, somewhat, 2=yes). Scores on this measure will be presented as means of all 4 items (range 0-2), where higher scores indicate higher recovery capital.
Experience of Support (Based on SAMHSA's definition of peer support) | Baseline, 1, 3, 6, and 12 months
  In conceptualizing and evaluating peer support services, SAMHSA (Substance Abuse and Mental Health Services Administration) distinguishes between four types of support: emotional, informational, instrumental, and affiliation support. To capture to what degree study participants experienced receiving these types of support, our study team created a 4-item self-report scale: (1) "I have experienced caring.";(2) "I have gained knowledge to help me reach my goals (e.g., wellness seminar, job training, parenting class, etc.)"; (3) "I have received concrete assistance to help me accomplish tasks (e.g., childcare, transportation, help accessing community health and social services)"; and (4) "I have felt a sense of belonging through shared activities with others." Each item is rated on a 4-point scale (3="Yes, a lot", 2="Yes, somewhat", 1="No, not really", 0="No, not at all"). Scores are averaged (range 0-3), where higher scores indicate higher levels of support.
The Brief Assessment of Recovery Capital (BARC-10) | Baseline, 1, 3, 6, and 12 months
  The Brief Assessment of Recovery Capital (BARC-10) is a 10-item self-report measure that is a short form of the 50-item Assessment of Recovery Capital (ARC) scale. Participants are asked to respond to each statement using a 6-point Likert scale ranging from 1 (="strongly disagree") to 6 (= "strongly agree"). The participant's response is then recorded and entered as a binary response option (agree = 1 / disagree = 0). The total score is the sum of all items that can range from 0 to 10, where higher scores indicate greater levels of recovery capital.
Participation in Recovery Support Services | Baseline, 1, 3, 6, and 12 months
  Participation in Recovery Support Services is a 3-item self-report questionnaire created by the investigators that assesses the participant's engagement (yes/no; if yes, how many days in the past 30 days) with a variety of recovery support services including mutual help organizations (e.g., Alcoholics Anonymous, Celebrate Recovery) and community recovery support services (e.g., recovery housing, recovery community centers). Answers will be summarized descriptively (% yes for listed mutual help organizations or recovery support services).
The Generalized Anxiety Disorder Screener (GAD-7) | Baseline, 1, 3, 6, and 12 months
  The Generalized Anxiety Disorder Screener (GAD-7) is a 7-item self-report scale that is used to assess the severity of generalized anxiety within participants over the previous 2-week period (e.g., "Feeling nervous, anxious or on edge."). Participants answer each item on a 4-point Likert scale ranging from 0 (= not at all) to 3 (= nearly every day). Scores are summed to a total score that can range from 0 to 21, where higher scores indicate more severe anxiety.
The Patient Health Questionnaire for Depression (PHQ-8) | Baseline, 1, 3, 6, and 12 months
  The Patient Health Questionnaire for Depression (PHQ-8) is an 8-item self-report measure used to assess participants' depression severity over the prior 2-week period (e.g., "Feeling down, depressed, or hopeless"). Participants answer each item on a 4-point Likert scale ranging from 0 = "Not at all (0 to 1 day)" to 3 = "Nearly every day (12-14 days)." Items are summed to form a total score that can range from 0 to 24, where higher scores indicate greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Hoeppner, Ph.D., M.S., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide de-identified IPD related to the aims, baseline demographics, and outcomes described in this study record to interested individuals one year following achievement of the aims of the project (i.e., publication of the main outcome papers). Data sharing will be contingent on meeting all institutional regulations for data use agreements and on receiving evidence of the recipient's institution's IRB approval for planned analyses of the data. The investigator team will be available to address queries.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will provide de-identified data from this project to interested individuals for one year following achievement of the aims of the project (i.e., publication of the main outcome papers).
Access Criteria: Data sharing will be contingent on meeting all institutional regulations for data use agreements and on receiving evidence of the recipient's institution's IRB approval for planned analyses of the data. Interested parties requesting data will receive the requested data needed to execute their analysis plan in accordance with these approvals. The IPD will be provided in digital format with clear labels for all variables, will be de-identified before it is shared, and will be released directly by the investigators to the recipients with secure data transfer.
  Regarding supporting information, the final version of the study protocol (including the statistical analysis plan (SAP)) and the final version of the Informed Consent Form (ICF) will be made publicly available in this clinicaltrials.gov record. Additional supporting information, including analytic code, will be made available upon a specific request to the investigative team.